CLINICAL TRIAL: NCT01189045
Title: Beyond VO2peak: Understanding Exercise-induced Changes in Cardiovascular Function After Stroke
Brief Title: Understanding Changes in Heart Function After Exercise in People With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-00735
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Rehabilitation; Risk factors
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Program (Experimental): The Aerobic Program will be the Experimental arm of this trial, where a structured, progressive aerobic exercise will be conducted in a class format
  Interventions: Behavioral: Aerobic Exercise Program
- Balance and Flexibility Program (Active Comparator): The Balance and Flexibility Program will be a non-aerobic intervention that will act as an Active Comparator. Stretching, balance exercises, yoga- or Tai Chi-style classes will be conducted.
  Interventions: Behavioral: Non-aerobic Exercise Program

INTERVENTIONS:
Behavioral: Aerobic Exercise Program — The AEROBIC PROGRAM will be the Experimental arm of this trial. It will be a structured, progressive aerobic training program that will be 6 months in duration. Classes will be held 3 times / week, for 1 hour / session.
  Arms: Aerobic Program
Behavioral: Non-aerobic Exercise Program — The BALANCE AND FLEXIBILITY (non-aerobic) PROGRAM will be the Active Comparator arm of this trial. It will be comprised of upper and lower body stretching, or balance activities, yoga- or Tai Chi-style classes. This program will be 6 months in duration. Classes will be held 3 times / week, for 1 hour / session.
  Arms: Balance and Flexibility Program

SUMMARY:
Little is known about how exercise can affect heart function in stroke survivors.

This study will look at changes in cardiovascular fitness and function after 6 months of exercise. Volunteers will be tested before and after the program and again 2 months later to measure the effects on stroke risk factors, fitness level and flexibility of the arteries. Blood tests will measure cholesterol levels and other signs of inflammation.

This study will help us better understand how exercise after stroke can improve heart function and heart health, and ultimately help in lowering future stroke risk.

DETAILED DESCRIPTION:
Purpose

To determine the effects of aerobic exercise after stroke on cardiorespiratory fitness, cardiovascular function, stroke risk factors, walking and health-related quality of life. This study will also examine the retention of these effects after the exercise program ends.

Methods

A randomized controlled study design will be used. Sixty participants will be randomized to participate in one of 2 treatment arms (6 months duration, 3 days / week, 1 hour / session):

1. BALANCE AND FLEXIBILITY (non-aerobic) PROGRAM will be comprised of individualized upper and lower body stretching, or balance activities, yoga- or Tai Chi-style classes.
2. AEROBIC PROGRAM will be comprised of a structured, progressive aerobic training program.

Participants will be evaluated at 3 time points - baseline (0 months), post-intervention (6 months) and follow up (8 months) - for stroke risk factors, cardiorespiratory fitness, arterial stiffness, echocardiography measures, inflammatory biomarkers, ambulatory capacity and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years old
* Has experienced a stroke
* At least 12 months post-stroke
* Able to stand independently
* Able to walk at least 5 metres (assisted devices and guarded supervision is permitted)

Exclusion Criteria:

* Stroke of non-cardiogenic origin (aneurysm, tumour)
* Actively engaged in other stroke rehabilitation services
* Class C or D American Heart Association Risk Criteria (uncontrolled arrhythmias)
* Resting blood pressure > 160/100 mmHg
* Significant musculoskeletal problems (rheumatoid arthritis) or other neurological conditions (e.g. Parkinson's)
* Has a pacemaker
* Pain or other co-morbidities (e.g. unclipped aneurysms, uncontrolled seizures etc.) which would preclude participation
* Behavioural issues that would limit participation in exercise

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Stroke risk factors (blood pressure, heart rate, lipid profiles, glucose metabolism), cardiorespiratory fitness | assessed at baseline (0 months), post-program (6 months) and follow up (8 months)

SECONDARY OUTCOMES:
Arterial stiffness and inflammatory biomarkers | assessed at 0, 6 and 8 months
Echocardiography measures | assessed at 0 and 6 months
Ambulatory capacity and health related quality of life | assessed at 0, 6 and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, PhD, Principal Investigator — The University of British Columbia - Vancouver Coastal Health Research Institute; Penelope Brasher, PhD, Study Director — Vancover General Hospital; Andrei Krassioukov, MD, PhD, Study Director — University of British Columbia; Kenneth Madden, MD, Study Director — University of British Columbia; Ada Tang, Study Director — University of British Columbia; Teresa Tsang, MD, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia